CLINICAL TRIAL: NCT02546960
Title: Randomized, Double-blind, Placebo-controlled, Multicenter Phase 2 Study in Healthy Adults to Evaluate the Safety and Immunogenicity of Different Doses of JNJ-63871860
Brief Title: A Study in Healthy Adults to Evaluate the Safety and Immunogenicity of Different Doses of JNJ-63871860
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CR107946; 63871860BAC2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Healthy
Keywords: Healthy; JNJ-63871860; ExPEC4V

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (6):
- ExPEC4V (4 : 4 : 4 : 4) (Experimental): Participants will be stratified according to their age in 2 groups >=18 to <50 years and >=50 years. Part 1: In age group >= 18 to <50 years, participants will receive single vaccination of ExPEC4V dose (4 : 4 : 4 : 4) as an intramuscular (i.m) injection into deltoid muscle. The ExPEC4V doses contain polysaccharide antigen (in microgram [mcg]) from the ExPEC serotypes O1A, O2, O6A, and O25B. Participants in >=50 years group will be enrolled in stepwise,dose-escalating procedure. In step 1, lowest dose of ExPEC4V (4:4:4:4) or Placebo will be given, in step 2 either of 2 medium doses of ExPEC4V or placebo and in step 3, either of 2 highest doses of ExPEC4V or placebo. Participants will be enrolled into subsequent steps only if vaccination in previous steps is deemed safe based on review of safety data by the IDMC. Participants will be enrolled into Part 2 only if vaccination in Part 1 is deemed safe based on the review of safety data through Day 8 by the IDMC.
  Interventions: Biological: ExPEC4V (4 : 4 : 4 : 4); Drug: Placebo
- ExPEC4V (4 : 4 : 4 : 8) (Experimental): Participants will be stratified according to their age in 2 groups >=18 to <50 years and >=50 years. Part 1: In age group >= 18 to <50 years, participants will receive single vaccination of ExPEC4V dose (4 : 4 : 4 : 8) as an i.m injection into deltoid muscle. The ExPEC4V doses contain polysaccharide antigen (in mcg) from the ExPEC serotypes O1A, O2, O6A, and O25B. Participants in >=50 years group will be enrolled in stepwise,dose-escalating procedure. In step 1, lowest dose of ExPEC4V or Placebo will be given, in step 2 either of 2 medium doses (4 : 4 : 4 : 8/8 : 8 : 8 : 8) of ExPEC4V or placebo and in step 3, either of 2 highest doses of ExPEC4V or placebo. Participants will be enrolled into subsequent steps only if vaccination in previous steps is deemed safe based on review of safety data by the IDMC. Participants will be enrolled into Part 2 only if vaccination in Part 1 is deemed safe based on the review of safety data through Day 8 by the IDMC.
  Interventions: Biological: ExPEC4V (4 : 4 : 4 : 8); Drug: Placebo
- ExPEC4V (8 : 8 : 8 : 8) (Experimental): Participants will be stratified according to their age in 2 groups >=18 to <50 years and >=50 years. Part 1: In age group >= 18 to <50 years, participants will receive single vaccination of ExPEC4V dose (8 : 8 : 8 : 8) as an i.m injection into deltoid muscle. The ExPEC4V doses contain polysaccharide antigen (in mcg) from the ExPEC serotypes O1A, O2, O6A, and O25B. Participants in >=50 years group will be enrolled in stepwise,dose-escalating procedure. In step 1, lowest dose of ExPEC4V or Placebo will be given, in step 2 either of 2 medium doses (4 : 4 : 4 : 8/8 : 8 : 8 : 8) of ExPEC4V or placebo and in step 3, either of 2 highest doses of ExPEC4V or placebo. Participants will be enrolled into subsequent steps only if vaccination in previous steps is deemed safe based on review of safety data by the IDMC. Participants will be enrolled into Part 2 only if vaccination in Part 1 is deemed safe based on the review of safety data through Day 8 by the IDMC.
  Interventions: Biological: ExPEC4V (8 : 8 : 8 : 8); Drug: Placebo
- ExPEC4V (8 : 8 : 8 : 16) (Experimental): Participants will be stratified according to their age in 2 groups >=18 to <50 years and >=50 years. Part 1: In age group >= 18 to <50 years, participants will receive single vaccination of ExPEC4V dose (8 : 8 : 8 : 16) as an i.m injection into deltoid muscle. The ExPEC4V doses contain polysaccharide antigen (in mcg) from the ExPEC serotypes O1A, O2, O6A, and O25B. Participants in >=50 years group will be enrolled in stepwise,dose-escalating procedure. In step 1, lowest dose of ExPEC4V or Placebo will be given, in step 2 either of 2 medium doses of ExPEC4V or placebo and in step 3, either of 2 highest doses (8 : 8 : 8 : 16/16 : 16 : 16 : 16) of ExPEC4V or placebo. Participants will be enrolled into subsequent steps only if vaccination in previous steps is deemed safe based on review of safety data by the IDMC. Participants will be enrolled into Part 2 only if vaccination in Part 1 is deemed safe based on the review of safety data through Day 8 by the IDMC.
  Interventions: Biological: ExPEC4V (8 : 8 : 8 : 16); Drug: Placebo
- ExPEC4V (16 : 16 : 16 : 16) (Experimental): Participants will be stratified according to their age in 2 groups >=18 to <50 years and >=50 years. Part 1: In age group >= 18 to <50 years, participants will receive single vaccination of ExPEC4V dose (16 : 16 : 16 : 16) as an i.m injection into deltoid muscle. The ExPEC4V doses contain polysaccharide antigen (in mcg) from the ExPEC serotypes O1A, O2, O6A, and O25B. Participants in >=50 years group will be enrolled in stepwise,dose-escalating procedure. In step 1, lowest dose of ExPEC4V or Placebo will be given, in step 2 either of 2 medium doses of ExPEC4V or placebo and in step 3, either of 2 highest doses (8 : 8 : 8 : 16/16 : 16 : 16 : 16) of ExPEC4V or placebo. Participants will be enrolled into subsequent steps only if vaccination in previous steps is deemed safe based on review of safety data by the IDMC. Participants will be enrolled into Part 2 only if vaccination in Part 1 is deemed safe based on the review of safety data through Day 8 by the IDMC.
  Interventions: Biological: ExPEC4V (16 : 16 : 16 : 16); Drug: Placebo
- Placebo (Placebo Comparator): Participants will be stratified according to their age in 2 groups >= 18 to <50 years and >=50 years. Part 1: Participants will receive matching placebo to ExPEC4V as an intramuscular injection into the deltoid muscle. Participants will be enrolled into Part 2 only if vaccination in Part 1 is deemed safe and well tolerated based on the review of safety data through Day 8 by the IDMC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: ExPEC4V (4 : 4 : 4 : 4) — Participants will receive single vaccination of ExPEC4V dose (4 : 4 : 4 : 4) as an intramuscular (i.m) injection into deltoid muscle in part 1 (age groups >=18 to <50 years and >=50 years) and part 2 (based on review of safety data by the IDMC). The ExPEC4V doses contain polysaccharide antigen (in microgram [mcg]) from the ExPEC serotypes O1A, O2, O6A, and O25B.
  Other Names: JNJ-63871860
  Arms: ExPEC4V (4 : 4 : 4 : 4)
Biological: ExPEC4V (4 : 4 : 4 : 8) — Participants will receive single vaccination of ExPEC4V dose (4 : 4 : 4 : 8) as an i.m injection into deltoid muscle in part 1 (age groups >=18 to <50 years and >=50 years) and part 2 (based on review of safety data by the IDMC). The ExPEC4V doses contain polysaccharide antigen (in mcg) from the ExPEC serotypes O1A, O2, O6A, and O25B.
  Other Names: JNJ-63871860
  Arms: ExPEC4V (4 : 4 : 4 : 8)
Biological: ExPEC4V (8 : 8 : 8 : 8) — Participants will receive single vaccination of ExPEC4V dose (8 : 8 : 8 : 8) as an i.m injection into deltoid muscle in part 1 (age groups >=18 to <50 years and >=50 years) and part 2 (based on review of safety data by the IDMC). The ExPEC4V doses contain polysaccharide antigen (in mcg) from the ExPEC serotypes O1A, O2, O6A, and O25B.
  Other Names: JNJ-63871860
  Arms: ExPEC4V (8 : 8 : 8 : 8)
Biological: ExPEC4V (8 : 8 : 8 : 16) — Participants will receive single vaccination of ExPEC4V dose (8 : 8 : 8 : 16) as an i.m injection into deltoid muscle in part 1 (age groups >=18 to <50 years and >=50 years) and part 2 (based on review of safety data by the IDMC). The ExPEC4V doses contain polysaccharide antigen (in mcg) from the ExPEC serotypes O1A, O2, O6A, and O25B.
  Other Names: JNJ-63871860
  Arms: ExPEC4V (8 : 8 : 8 : 16)
Biological: ExPEC4V (16 : 16 : 16 : 16) — Participants will receive single vaccination of ExPEC4V dose (16 : 16 : 16 : 16) as an i.m injection into deltoid muscle in part 1 (age groups >=18 to <50 years and >=50 years) and part 2 (based on review of safety data by the IDMC). The ExPEC4V doses contain polysaccharide antigen (in mcg) from the ExPEC serotypes O1A, O2, O6A, and O25B.
  Other Names: JNJ-63871860
  Arms: ExPEC4V (16 : 16 : 16 : 16)
Drug: Placebo — Participants will receive matching placebo (Tris-buffered saline) to ExPEC4V.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability of different doses of JNJ-63871860 (ExPEC4V) in participants greater than or equal to (>=)18 years of age and to evaluate the dose-dependent immunogenicity of ExPEC as measured by enzyme-linked immunosorbent assay (ELISA).

DETAILED DESCRIPTION:
This is a Phase 2, double-blind (neither the researchers nor the participants know what treatment the participant is receiving), randomized (study medication assigned to participants by chance), placebo-controlled (an inactive substance; a pretend treatment [with no drug in it] that is compared in a clinical trial with a drug to test if the drug has a real effect), parallel group, multicenter (when more than one hospital work on a medical research study) study, with a single-blind, long-term follow-up to Year 3. The study will be split into 2 phases, a double-blind phase with screening (Day -12 to Day 1), Vaccination (Day 1) and Safety and Immunogenicity Follow-up (Day 1 up to Day 360), and a single-blind long-term follow-up phase thereafter until Year 3 for participants in placebo and two ExPEC4V dose groups selected based on the primary (Day 30) analysis. Participants will be stratified in 2 age groups (>=18 to less than [<] 50 years and >=50 years) and in each dosing group in each stratum randomized to a single vaccination with 1 of 5 doses of ExPEC4V or placebo. The duration of the double-blind phase (from randomization/vaccination) will be approximately 360 days for placebo participants and participants in the dose group selected based on the primary analysis, and approximately 180 days for the participants in the other groups. The duration of the single-blind long-term follow-up phase will be approximately 2 years after the double-blind phase for placebo participants and participants in the selected dose group. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be in stable health. Participants may have underlying illnesses such as hypertension, diabetes, ischemic heart disease, hyperlipoproteinemia, or hypothyroidism, as long as their symptoms/signs are medically controlled. If they are on medication for a condition, the medication dose must have been stable for at least 12 weeks preceding vaccination and is expected to remain stable for the duration of the study
* Participant must meet the protocol defined laboratory criteria within 12 days before Day 1
* Participant must be able to attend all scheduled visits and to comply with all study procedures
* Participant must have a body mass index (BMI) of less than or equal to (<=) 35 kilogram per square meter (kg/m^2)
* A woman of childbearing potential must have a negative urine pregnancy test on Day 1 before vaccination

Exclusion Criteria:

* Participant is a woman who is pregnant, breast-feeding, or has a positive urine pregnancy test on Day 1 before vaccination, or is planning to become pregnant 3 months after study vaccine administration or within 3 months after study vaccine administration, or subject is a man who plans to father a child while enrolled in this study or within 3 months after study vaccine administration
* Participant has an acute illness, acute infection, or fever (body temperature greater than or equal to [>=] 38 degree Celsius)
* Participant has a serious chronic disorder, including severe chronic obstructive pulmonary disease or clinically significant congestive heart failure, requirement for supplemental oxygen, end stage renal disease with or without dialysis, clinically unstable cardiac disease, or has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (example compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Participant has a history of neoplastic disease (excluding non-melanoma skin cancer that was successfully treated) within the past 5 years or a history of any hematological malignancy
* Participant has known or suspected congenital or acquired immunodeficiency (including leukemia, HIV seropositivity), has received immunosuppressive therapy (such as anti-cancer chemotherapy, radiation therapy or cytotoxic drugs), within the preceding 6 months; or long-term systemic corticosteroid therapy [prednisone or equivalent for more than 2 consecutive weeks within the past 3 months]), or has chronic active hepatitis B or hepatitis C infection, documented by hepatitis B surface antigen and hepatitis C antibody, respectively

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 848 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2016-09-12 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local Adverse Events (AEs) | up to Day 8
  Solicited AEs are precisely defined events that participants are specifically asked about and which are noted by participants through the electronic Subject Diary. Solicited Local AEs: Participants will be instructed on how to note occurrences of pain/tenderness, erythema, and induration/swelling at the injection site daily for 8 days postvaccination (day of vaccination and the subsequent 7 days) in the electronic Subject Diary. Participants will be instructed on how to measure (using the ruler supplied) and record erythema and induration.
Number of Participants with Solicited Systemic AEs | up to Day 8
  Solicited AEs are precisely defined events that participants are specifically asked about and which are noted by participants through the electronic Subject Diary. Solicited Systemic AEs: Participants will be instructed on how to note daily symptoms in the electronic Subject Diary for 8 days post vaccination (day of vaccination and the subsequent 7 days) of the following systemic events: fever, headache, fatigue, malaise, nausea, and myalgia.
Number of Participants with Unsolicited AEs | Up to Day 30
Number of Participants with Serious Adverse Events (SAE's) | Until 360 days post vaccination
  An SAE is any adverse event that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Dose-dependent Immunogenicity of ExPEC4V on Day 15 (ELISA) | Day 15
  Dose-dependent immunogenicity will be measured by enzyme-linked immunosorbent assay (ELISA) on day 15 in participants with >=18 years of age. Immunoglobulin G (IgG) antibody levels elicited by the vaccine will be measured by ELISA.
Long-Term Immunogenicity of ExPEC4V Dose Selected for Further Clinical Development (ELISA) | Year 2 and 3
  Evaluation of the immunogenicity of a single vaccination with the ExPEC4V dose selected for further clinical development based on the primary analysis, as measured by ELISA.

SECONDARY OUTCOMES:
Dose-dependent Immunogenicity of ExPEC4V on Day 15 (Opsonophagocytic Killing [OPK] Assay) | Day 15
  Dose-dependent immunogenicity will be measured by opsonophagocytic killing (OPK) assay on day 15 in participants with >=18 years of age. Specific functional antibacterial antibodies will be measured by OPK.
Correlation Between ELISA (total antibody) and OPK (functional antibody) Serum Titers | Day 15
Dose-dependent Immunogenicity of ExPEC4V on Day 30 (ELISA) | Day 30
  Dose-dependent immunogenicity will be measured by ELISA on day 30 in participants with >=18 years of age. IgG antibody levels elicited by the vaccine will be measured by ELISA.
Immunogenicity of ExPEC4V Dose Selected for Further Clinical Development (ELISA) | Day 180 and 360
  The immunogenicity of the ExPEC4V dose selected for further clinical development based on the interim analysis, as measured by ELISA will be evaluated. IgG antibody levels elicited by the vaccine will be measured by ELISA.
Immunogenicity of ExPEC4V Dose Selected for Further Clinical Development (OPK) | Days 30, 180, and 360
  The immunogenicity of the ExPEC4V dose selected for further clinical development based on the interim analysis, as measured by OPK assay will be evaluated. Specific functional antibacterial antibodies will be measured by OPK.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Mesa, Arizona
  - Hollywood, Florida
  - Leesburg, Florida
  - Miami, Florida
  - Boise, Idaho
  - Wichita, Kansas
  - Bardstown, Kentucky
  - Baltimore, Maryland
  - Saint Paul, Minnesota
  - Kansas City, Missouri
  - Las Vegas, Nevada
  - Cary, North Carolina
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Knoxville, Tennessee
  - Austin, Texas
  - Houston, Texas

REFERENCES:
- [Derived] Frenck RW Jr, Ervin J, Chu L, Abbanat D, Spiessens B, Go O, Haazen W, van den Dobbelsteen G, Poolman J, Thoelen S, Ibarra de Palacios P. Safety and immunogenicity of a vaccine for extra-intestinal pathogenic Escherichia coli (ESTELLA): a phase 2 randomised controlled trial. Lancet Infect Dis. 2019 Jun;19(6):631-640. doi: 10.1016/S1473-3099(18)30803-X. Epub 2019 May 9. PMID 31079947